CLINICAL TRIAL: NCT02940925
Title: TPC vs PF as Induction Chemotherapy Combined With CCRT for Stage IVa-b Nasopharyngeal Carcinoma, a Prospective,Parallel, Randomized, Open Labeled, Multicenter Phase III Clinical Trial
Brief Title: TPC vs PF as Induction Chemotherapy Combined With CCRT for Stage IVa-b Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, XIANG YANQUN, PROFESSOR, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20160049
Record Dates: First submitted 2016-09-21; First posted 2016-10-21 (Estimated); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; induction chemotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Paclitaxel; Cisplatin; Capecitabine; Fluorouracil

STUDY DESIGN:
Intervention Model Description: Experimental: Drug: Taxol,cisplatin and capecitabine Active Comparator: Drug: Cisplatin and 5-Fluorouracil
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug: Taxol,cisplatin and capecitabine (Experimental): Taxol, cisplatin and capecitabine as induction chemotherapy (IC) combined with cisplatin concurrent chemoradiotherapy with intensity modulated radiation therapy |(CCRT).
  Interventions: Other: Drug: Taxol,cisplatin and capecitabine
- Drug: Cisplatin and 5-Fluorouracil (Active Comparator): Cisplatin and 5-Fluorouracil as induction chemotherapy combined with cisplatin concurrent chemoradiotherapy with intensity modulated radiation therapy.
  Interventions: Other: Drug: Cisplatin and 5-Fluorouracil

INTERVENTIONS:
Other: Drug: Taxol,cisplatin and capecitabine — Taxol, cisplatin and capecitabine as induction chemotherapy combined with cisplatin concurrent chemoradiotherapy with intensity modulated radiation therapy.
  Arms: Drug: Taxol,cisplatin and capecitabine
Other: Drug: Cisplatin and 5-Fluorouracil — Cisplatin and 5-Fluorouracil as induction chemotherapy combined with cisplatin concurrent chemoradiotherapy with intensity modulated radiation therapy.
  Arms: Drug: Cisplatin and 5-Fluorouracil

SUMMARY:
The purpose of this study is to compare the survival and toxicity of TPC (TAXOL, DDP AND CAPECITABINE ) VS PF (cisplatin and 5-Fluorouracil) as induction chemotherapy combined with concurrent chemoradiotherapy (CCRT) for stage IVa-b nasopharyngeal carcinoma patients in endemic area.

DETAILED DESCRIPTION:
This is a prospective, parallel, randomized, open labeled, multicenter phase III clinical trial to compare the survival and toxicity of TPC VS PF as induction chemotherapy combined with CCRT for stage IVa-b nasopharyngeal carcinoma patients in endemic area.The primary endpoint is failure free survival (FFS）.The secondary endpoints are overall survival(OS）,progression-free survival（PFS）, local-regionally relapse free survival(LRFS), distant metastasis free survival（DMFS)and toxicities.

ELIGIBILITY:
Inclusion Criteria:

* WHO II or III pathological type
* stage Ⅳa or Ⅳb (UICC 7th edition)
* no anticancer treatment before
* no malignant history
* both gender, 18-60 years old
* enough liver function: TBIL≤ULN；AST/ALT≤2.5×ULN；ALP≤5×ULN
* enough kidney function: Clcr≥80 mL/min
* enough hemo: ANC≥2×109/L, PLT≥100×109/L and HB≥9g/dL
* no sever heart, lung disfunction
* PS≤2

Exclusion Criteria:

* previous anticancer treatment
* distant metastasis
* pregnant or breasting female
* can not access to followup
* enrolled in other therapeutic clinical trial
* sever infection and internal disease
* sever disfunction of heart, lung, kidney, liver, etc
* TBIL>ULN；AST/ALT>2.5×ULN；ALP>5×ULN
* with factors that will affect the administration, distribution,metabolism or evacuation.
* using immunosuppressive agents after organ transplantation
* other malignant history

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 241 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2021-08-28 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Failure-free survival calculated from randomisation to locoregional failure, distant failure, or death from any cause | up to 5 years

SECONDARY OUTCOMES:
Overall survival calculated from randomisation to death from any cause | up to 5 years
Progression free survival calculated from randomisation to disease progression or death from any cause | up to 5 years
Local-regionally relapse free survival calculated from randomisation to locoregional failure | up to 5 years
Distant metastasis free survival calculated from randomisation to distant failure | up to 5 years
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yanqun Xiang, Study Chair — Sun Yat-sen University; Taize Yuan, Principal Investigator — Cancer Center of Guangzhou medical school; Yunxiang He, Principal Investigator — Xiangya Hospital
Locations (1):
- SunYat-senU, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The diagnosis, treatment regimen, toxicity and followup data will be shared once every year through email, phone or meeting.

REFERENCES:
- [Background] Hui EP, Ma BB, Leung SF, King AD, Mo F, Kam MK, Yu BK, Chiu SK, Kwan WH, Ho R, Chan I, Ahuja AT, Zee BC, Chan AT. Randomized phase II trial of concurrent cisplatin-radiotherapy with or without neoadjuvant docetaxel and cisplatin in advanced nasopharyngeal carcinoma. J Clin Oncol. 2009 Jan 10;27(2):242-9. doi: 10.1200/JCO.2008.18.1545. Epub 2008 Dec 8. PMID 19064973
- [Background] Chan AT, Ma BB, Lo YM, Leung SF, Kwan WH, Hui EP, Mok TS, Kam M, Chan LS, Chiu SK, Yu KH, Cheung KY, Lai K, Lai M, Mo F, Yeo W, King A, Johnson PJ, Teo PM, Zee B. Phase II study of neoadjuvant carboplatin and paclitaxel followed by radiotherapy and concurrent cisplatin in patients with locoregionally advanced nasopharyngeal carcinoma: therapeutic monitoring with plasma Epstein-Barr virus DNA. J Clin Oncol. 2004 Aug 1;22(15):3053-60. doi: 10.1200/JCO.2004.05.178. PMID 15284255
- [Background] Vermorken JB, Remenar E, van Herpen C, Gorlia T, Mesia R, Degardin M, Stewart JS, Jelic S, Betka J, Preiss JH, van den Weyngaert D, Awada A, Cupissol D, Kienzer HR, Rey A, Desaunois I, Bernier J, Lefebvre JL; EORTC 24971/TAX 323 Study Group. Cisplatin, fluorouracil, and docetaxel in unresectable head and neck cancer. N Engl J Med. 2007 Oct 25;357(17):1695-704. doi: 10.1056/NEJMoa071028. PMID 17960012
- [Background] Lee AW, Ngan RK, Tung SY, Cheng A, Kwong DL, Lu TX, Chan AT, Chan LL, Yiu H, Ng WT, Wong F, Yuen KT, Yau S, Cheung FY, Chan OS, Choi H, Chappell R. Preliminary results of trial NPC-0501 evaluating the therapeutic gain by changing from concurrent-adjuvant to induction-concurrent chemoradiotherapy, changing from fluorouracil to capecitabine, and changing from conventional to accelerated radiotherapy fractionation in patients with locoregionally advanced nasopharyngeal carcinoma. Cancer. 2015 Apr 15;121(8):1328-38. doi: 10.1002/cncr.29208. Epub 2014 Dec 19. PMID 25529384
- [Background] Gao Y, Huang HQ, Bai B, Cai QC, Wang XX, Cai QQ. Treatment outcome of docetaxel, capecitabine and cisplatin regimen for patients with refractory and relapsed nasopharyngeal carcinoma who failed previous platinum-based chemotherapy. Expert Opin Pharmacother. 2014 Feb;15(2):163-71. doi: 10.1517/14656566.2014.866652. Epub 2013 Dec 3. PMID 24295173
- [Derived] Li WZ, Lv X, Hu D, Lv SH, Liu GY, Liang H, Ye YF, Yang W, Zhang HX, Yuan TZ, Wang DS, Lu N, Ke LR, Tang WB, Tong LH, Chen ZJ, Liu T, Cao KJ, Mo HY, Guo L, Zhao C, Chen MY, Chen QY, Huang PY, Sun R, Qiu F, Luo DH, Wang L, Hua YJ, Tang LQ, Qian CN, Mai HQ, Guo X, Xiang YQ, Xia WX. Effect of Induction Chemotherapy With Paclitaxel, Cisplatin, and Capecitabine vs Cisplatin and Fluorouracil on Failure-Free Survival for Patients With Stage IVA to IVB Nasopharyngeal Carcinoma: A Multicenter Phase 3 Randomized Clinical Trial. JAMA Oncol. 2022 May 1;8(5):706-714. doi: 10.1001/jamaoncol.2022.0122. PMID 35323856